CLINICAL TRIAL: NCT05659329
Title: A Retrospective Multicenter Study to Review the Use of Simplex High Viscosity Bone Cement in Primary Total Knee Arthroplasty
Brief Title: Retrospective Simplex High Viscosity (HV) Bone Cement Study
Status: Completed | Type: Observational
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 80
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-07

CONDITIONS: Arthritis Knee; Aseptic Loosening
Keywords: Bone Cement; Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Non-medicated Simplex HV: Retrospective observation of patients who have received a Triathlon Total Knee Replacement implanted with nonmedicated Simplex HV Bone Cement.
  Interventions: Device: Simplex HV/Gentamicin Simplex HV bone cement
- Gentamicin Simplex HV: Retrospective observation of patients who have received a Triathlon Total Knee Replacement implanted with Gentamicin Simplex HV Bone Cement.
  Interventions: Device: Simplex HV/Gentamicin Simplex HV bone cement

INTERVENTIONS:
Device: Simplex HV/Gentamicin Simplex HV bone cement — Simplex HV bone cement is a fast-setting acrylic resin for use in bone surgery.
  Simplex HV bone cement with Gentamicin is a fast setting acrylic resin with addition of gentamicin sulfate for use in bone surgery.
  Mixing two separate sterile components produces a ductile bone cement which, after hardening, fixes the implant and transfers stresses produced during movement evenly to the bone.

SUMMARY:
This study is a retrospective multicenter study to review the use of Simplex High Viscosity Bone Cement in Primary Total Knee Arthroplasty

DETAILED DESCRIPTION:
This study is a retrospective investigation of subjects who have received primary Triathlon Total Knee Arthroplasty inserted with Simplex High Viscosity (HV) Cement to evaluate the success rate defined as absence of revision for aseptic loosening of components at two years postoperative.

ELIGIBILITY:
Inclusion Criteria:

* The Patient is age 18 or over at time of study device implantation
* Patients who have undergone primary Triathlon Total Knee Arthroplasty in which Simplex HV/Simplex HV Gentamicin was indicated for fixation and used on label
* Patients who have been followed for at least 24 months postoperatively

Exclusion Criteria:

* Patients who have undergone revision surgery
* Patients who have undergone bilateral Knee Arthroplasty
* Patients contraindicated for either the devices implanted, or the cement used, according to medical history review and instructions for use
* Patient has a cementless tibial baseplate.
* Patient has an active or suspected latent infection in or about the affected knee joint
* Patient has muscle loss or neuromuscular impairment in the affected limb that would create an unjustifiable risk
* Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days)
* Patient has a known hypersensitivity to any of the cements constituents or in patients with severe renal failure
* Patient is a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all non-censored subjects who have received the Triathlon total knee system cemented with Simplex HV and are available for objective analysis.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Toms, Prof., Principal Investigator — PEOC Royal Devon & Exeter Hospital; Matthew Hepinstall, MD, Principal Investigator — Department of Orthopedic Surgery NYU Langone Health

IPD SHARING:
Plan to Share IPD: No
not planned

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a retrospective study with planned 100 subjects per group. Recruitment was stopped in the Non-medicated Simplex HV group with 97 subjects because there were no additional eligible subjects.
Pre-assignment Details: In the non-medicated Simplex HV group further three of the 97 subjects were excluded after enrollment as two subjects did not receive the study device and one subject met an exclusion criterion (Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days))
Groups:
- Non-medicated Simplex HV: Retrospective observation of patients who have received a Triathlon Total Knee Replacement implanted with nonmedicated Simplex HV Bone Cement.
  Simplex HV Bone Cement is a fast-setting acrylic resin for use in bone surgery. Mixing the two separate sterile components produces a ductile bone cement which, after hardening, fixes the implant and transfers stresses produced during movement evenly to the bone.
- Gentamicin Simplex HV: Retrospective observation of patients who have received a Triathlon Total Knee Replacement implanted with Gentamycin Simplex HV Bone Cement.
  Gentamicin Simplex HV Bone Cement is a fast-setting acrylic resin with addition of gentamicin sulfate for use in bone surgery. Mixing the two separate sterile components produces a ductile bone cement which, after hardening, fixes the implant and transfers stresses produced during movement evenly to the bone.
Period: Overall Study
Arm/Group | Non-medicated Simplex HV | Gentamicin Simplex HV
Started | 95 | 101
Completed | 95 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gentamicin Simplex HV: Retrospective observation of patients who have received a Triathlon Total Knee Replacement implanted with Gentamycin Simplex HV Bone Cement.
  Simplex HV Bone Cement with Gentamicin is a fast-setting acrylic resin with addition of gentamicin sulfate for use in bone surgery. Mixing the two separate sterile components produces a ductile bone cement which, after hardening, fixes the implant and transfers stresses produced during movement evenly to the bone.
- Total: Total of all reporting groups
Arm/Group | Non-medicated Simplex HV | Gentamicin Simplex HV | Total
Number analyzed (Participants) | 95 | 101 | 196
Age, Customized [Mean (Standard Deviation); unit: years] | 66 (8.84) | 71.8 (7.83) | 68.97 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 58 | 123
  Male | 30 | 43 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 95 | 0 | 95
  United Kingdom | 0 | 101 | 101
Height cm [Mean (Standard Deviation); unit: centimeter] — Population: In the Simplex HV Gentamicin group, for some subjects height was not available in retrospective data collection.
  centimeter | 165 (10.17) | 166 (9.24) | 165.4 (9.7)
Weight kg [Mean (Standard Deviation); unit: kilogram] | 91.0 (19.65) | 83.4 (14.82) | 87.1 (17.71)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.3 (5.94) | 30.5 (4.73) | 31.87 (5.53)
Operative side [Count of Participants; unit: Participants]
  Left side | 47 | 44 | 91
  Right side | 48 | 57 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Application of Bone Cement
Description: A successful application is defined as absence of revision of Triathlon Total Knee components cemented with Simplex high viscosity bone cement (Simplex HV) within outcome measure timeframe.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Gentamicin Simplex HV: Retrospective observation of patients who have received a Triathlon Total Knee Replacement implanted with Gentamicin Simplex HV Bone Cement.
  Gentamicin Simplex HV Bone Cement is a fast-setting acrylic resin with addition of gentamicin sulfate for use in bone surgery. Mixing the two separate sterile components produces a ductile bone cement which, after hardening, fixes the implant and transfers stresses produced during movement evenly to the bone.
Arm/Group | Non-medicated Simplex HV | Gentamicin Simplex HV
Number analyzed (Participants) | 95 | 101
Participants | 95 | 101

2. Secondary Outcome: Knee Society Score (KSS) Pain Motion Score: Range of Motion
Description: The Knee range of motion (ROM) is a parameter which is calculating the range of knee extension (the ability to straighten the leg) and knee flexion (ability to bend the leg). A normal range is from 0º extension (completely straight leg) to 130º flexion (fully flexed leg).
Time Frame: pre-op, 2 years, 5 years (optional)
Population: The retrospective study approach did not allow for full KSS data collection. Range of motion data available were collected for analysis.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Non-medicated Simplex HV | Gentamicin Simplex HV
Number analyzed (Participants) | 90 | 26
degrees
  Pre-op Range of motion (ROM) | 108.59 (12.74) | 101.16 (14.19)
  2 years ROM: number analyzed (Participants) | 82 | 8
  2 years ROM | 110.48 (12.48) | 110.32 (11.40)
  5 years ROM: number analyzed (Participants) | 49 | 8
  5 years ROM | 113.37 (13.35) | 114.81 (8.74)

3. Secondary Outcome: KSS Pain Motion Score: Pain
Description: This section shows a five-level pain measurement from "no pain" to "severe pain" reported by the subjects.
Time Frame: Pre-operative, 2 years, 5 years (optional)
Population: The retrospective study approach did not allow for full KSS data collection. Pain data available were collected for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Gentamycin Simplex HV: Retrospective observation of patients who have received a Triathlon Total Knee Replacement implanted with Gentamycin Simplex HV Bone Cement.
  Gentamicin Simplex HV Bone Cement is a fast-setting acrylic resin with addition of gentamicin sulfate for use in bone surgery.
  Mixing the two separate sterile components produces a ductile bone cement which, after hardening, fixes the implant and transfers stresses produced during movement evenly to the bone.
Arm/Group | Non-medicated Simplex HV | Gentamycin Simplex HV
Number analyzed (Participants) | 90 | 26
Participants
  Pre-operative Pain: No pain | 0 | 1
  Pre-operative Pain: Mild or occasional pain | 11 | 0
  Pre-operative Pain: Moderate continual pain | 34 | 6
  Pre-operative Pain: Moderate occasional pain | 24 | 1
  Pre-operative Pain: Severe pain | 21 | 18
  Pain at 2 years: number analyzed (Participants) | 82 | 8
  Pain at 2 years: No pain | 49 | 2
  Pain at 2 years: Mild or occasional pain | 26 | 5
  Pain at 2 years: Moderate continual pain | 3 | 0
  Pain at 2 years: Moderate occasional pain | 4 | 0
  Pain at 2 years: Severe pain | 0 | 1
  Pain at 5 years: number analyzed (Participants) | 49 | 8
  Pain at 5 years: No pain | 29 | 6
  Pain at 5 years: Mild or occasional pain | 17 | 2
  Pain at 5 years: Moderate continual pain | 1 | 0
  Pain at 5 years: Moderate occasional pain | 2 | 0
  Pain at 5 years: Severe pain | 0 | 0

4. Secondary Outcome: KSS Function Score: Walking Aids
Description: Pre- and postoperative use of walking aids
Time Frame: Pre-operative, 2 years, 5 years (optional)
Population: The retrospective study approach did not allow for full KSS data collection. Use of walking aids data available were collected for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-medicated Simplex HV | Gentamycin Simplex HV
Number analyzed (Participants) | 69 | 23
Participants
  Pre-operative walking aids use: Cane | 23 | 12
  Pre-operative walking aids use: Crutches, Walker, cannot walk/ wheelchair Crutches, Walker, cannot walk, wheelchair | 3 | 1
  Pre-operative walking aids use: Two canes, one crutch | 0 | 1
  Pre-operative walking aids use: None | 43 | 9
  Walking aids use at 2 years: number analyzed (Participants) | 67 | 2
  Walking aids use at 2 years: Cane | 13 | 0
  Walking aids use at 2 years: Crutches, Walker, cannot walk/ wheelchair Crutches, Walker, cannot walk, wheelchair | 2 | 0
  Walking aids use at 2 years: Two canes, one crutch | 0 | 0
  Walking aids use at 2 years: None | 52 | 2
  Walking aids use at 5 years: number analyzed (Participants) | 40 | 0
  Walking aids use at 5 years: Cane | 8 |
  Walking aids use at 5 years: Crutches, Walker, cannot walk/ wheelchair Crutches, Walker, cannot walk, wheelchair | 2 |
  Walking aids use at 5 years: Two canes, one crutch | 0 |
  Walking aids use at 5 years: None | 30 |

5. Secondary Outcome: KSS Function Score: Walking
Description: Pre- and post-operative walking ability
Time Frame: pre-operative, 2 years, 5 years (optional)
Population: The retrospective study approach did not allow for full KSS data collection. Walking ability data available were collected for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-medicated Simplex HV | Gentamycin Simplex HV
Number analyzed (Participants) | 52 | 24
Participants
  Pre-operative walking ability: Housebound | 1 | 0
  Pre-operative walking ability: Below 5 blocks (<500m/<1640 feet) | 48 | 13
  Pre-operative walking ability: 5-10 blocks (500m - 1000m/1640-3280 feet) | 0 | 7
  Pre-operative walking ability: Over 10 blocks (>1000m/>3280 feet) | 2 | 2
  Pre-operative walking ability: Unlimited | 1 | 2
  Walking ability at 2 years: number analyzed (Participants) | 24 | 3
  Walking ability at 2 years: Housebound | 2 | 0
  Walking ability at 2 years: Below 5 blocks (<500m/<1640 feet) | 2 | 0
  Walking ability at 2 years: 5-10 blocks (500m - 1000m/1640-3280 feet) | 0 | 0
  Walking ability at 2 years: Over 10 blocks (>1000m/>3280 feet) | 3 | 1
  Walking ability at 2 years: Unlimited | 17 | 2
  Walking ability at 5 years: number analyzed (Participants) | 16 | 3
  Walking ability at 5 years: Housebound | 0 | 0
  Walking ability at 5 years: Below 5 blocks (<500m/<1640 feet) | 1 | 0
  Walking ability at 5 years: 5-10 blocks (500m - 1000m/1640-3280 feet) | 2 | 1
  Walking ability at 5 years: Over 10 blocks (>1000m/>3280 feet) | 0 | 0
  Walking ability at 5 years: Unlimited | 13 | 2

6. Secondary Outcome: KSS Function Score: Stairs
Description: Pre-and postoperative ability of climbing stairs
Time Frame: Pre-operative, 2 years, 5 years (optional)
Population: The retrospective study approach did not allow for full KSS data collection. Stair climbing ability data available were collected for analysis of non-medicated Simplex HV only.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-medicated Simplex HV | Gentamycin Simplex HV
Number analyzed (Participants) | 36 | 0
Participants
  Pre-operative ability to climb stairs: Unable | 22 |
  Pre-operative ability to climb stairs: Up with rail/unable down | 0 |
  Pre-operative ability to climb stairs: Up and down with rail | 12 |
  Pre-operative ability to climb stairs: Normal up/down with rail | 2 |
  Pre-operative ability to climb stairs: Normal up and down | 0 |
  Ability to climb stairs at 2 years: number analyzed (Participants) | 18 | 0
  Ability to climb stairs at 2 years: Unable | 0 |
  Ability to climb stairs at 2 years: Up with rail/unable down | 0 |
  Ability to climb stairs at 2 years: Up and down with rail | 2 |
  Ability to climb stairs at 2 years: Normal up/down with rail | 1 |
  Ability to climb stairs at 2 years: Normal up and down | 15 |
  Ability to climb stairs at 5 years: number analyzed (Participants) | 17 | 0
  Ability to climb stairs at 5 years: Unable | 1 |
  Ability to climb stairs at 5 years: Up with rail/unable down | 0 |
  Ability to climb stairs at 5 years: Up and down with rail | 2 |
  Ability to climb stairs at 5 years: Normal up/down with rail | 1 |
  Ability to climb stairs at 5 years: Normal up and down | 13 |

7. Secondary Outcome: Oxford Knee Score (OKS) Results
Description: The OKS is a patient reported outcome measure that consists of 12 questions about an individual's level of function, activities of daily living and how they have been affected by pain over the preceding four weeks. On a scale between 0 and 48, low values indicate severe knee problems and high values indicate satisfactory joint function.
Time Frame: pre-op, 2 years, 5 years (optional)
Population: Due to the retrospective study approach, the site of the Non-medicated Simplex HV arm did not collect OKS data and therefore OKS data cannot be presented for this site, whereas the site for the Gentamicin Simplex HV arm did collect OKS data which are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-medicated Simplex HV | Gentamicin Simplex HV
Number analyzed (Participants) | 0 | 101
score on a scale
  pre-operative OKS |  | 18.96 (7.79)
  2 years OKS: number analyzed (Participants) | 0 | 57
  2 years OKS |  | 39.27 (7.92)
  5 years OKS: number analyzed (Participants) | 0 | 42
  5 years OKS |  | 39.38 (7.73)

8. Secondary Outcome: KSS Pain Motion Score: Stability
Description: This section shows number of patients with a minor knee ligament laxity. Antero-posterior (a/p) stability < 5 mm and medio-lateral (m/l) stability < 5° means mild increase in laxity compared to the contralateral knee.
Time Frame: pre-operative, 2 years, 5 years (optional)
Population: The retrospective study approach in the Non-medicated Simplex HV study arm did not allow for full KSS Stability data collection as not all data were collected at 2 and 5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-medicated Simplex HV | Gentamicin Simplex HV
Number analyzed (Participants) | 87 | 1
Participants
  preoperative a/p <5mm and m/l <5° stability | 87 | 1
  2 years a/p <5mm and m/l <5° stability: number analyzed (Participants) | 81 | 0
  2 years a/p <5mm and m/l <5° stability | 81 | 0
  5 years a/p <5mm and m/l <5° stability: number analyzed (Participants) | 52 | 0
  5 years a/p <5mm and m/l <5° stability | 52 | 0

ADVERSE EVENTS:
Time Frame: In this retrospective study adverse events were collected from time point of study related surgery up to 2 years.
Description: No difference to ClinicalTrials.gov definition.
Arm/Group | Non-medicated Simplex HV | Gentamicin Simplex HV
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/101
Serious Adverse Events (participants affected / at risk) | 10/95 | 21/101
Other Adverse Events (participants affected / at risk) | 18/95 | 9/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-medicated Simplex HV (N=95) | Gentamicin Simplex HV (N=101)
Non-operative (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Non-operative (Cardiac disorders) | 2 (2) | 2 (3)
Non-operative (Gastrointestinal disorders) | 1 (1) | 1 (1)
Non-operative (Immune system disorders) | 0 (0) | 1 (1)
Non-operative (Infections and infestations) | 1 (1) | 1 (1)
Non-operative (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Non-operative (Nervous system disorders) | 0 (0) | 1 (1)
Non-operative (Psychiatric disorders) | 1 (1) | 0 (0)
Non-operative (Renal and urinary disorders) | 1 (1) | 3 (3)
Non-operative (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Non-operative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Non-operative (Vascular disorders) | 0 (0) | 1 (1)
Non-operative (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Operative site (Surgical and medical procedures) | 0 (0) | 3 (3)
Operative site (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-medicated Simplex HV (N=95) | Gentamicin Simplex HV (N=101)
Operative site (Musculoskeletal and connective tissue disorders) | 18 (24) | 9 (9)

LIMITATIONS AND CAVEATS:
The retrospective study approach did not allow for full KSS data collection. Data available were collected for analysis. In the retrospective data collection of this study, for some subjects were either no data or 2 years, respective 5 years data available. 5 years data are not mandatorily a consecutive follow-up of the 2 years data of the same subject. OKS was available for one site only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT05659329/Prot_SAP_000.pdf